CLINICAL TRIAL: NCT01752920
Title: A Phase 1/2 Study of ARQ 087 in Adult Subjects With Advanced Solid Tumors With FGFR Genetic Alterations, Including Intrahepatic Cholangiocarcinoma With FGFR2 Gene Fusion
Brief Title: Phase 1/2 Study of Derazantinib (ARQ 087) in Adult Subjects With Advanced Solid Tumors With FGFR Genetic Alterations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 087-101
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
Keywords: FGFR; ARQ 087; Targeted therapy; Molecular therapy; Tyrosine kinase inhibitor; TKI; Receptor tyrosine kinase; RTK; Biomarker; Phase 1; Phase I; Solid tumor; Liver Cancer; Hepatobiliary carcinoma; Biliary tract cancer; Cholangiocarcinoma; Intrahepatic cholangiocarcinoma; FGFR inhibitor; Targeted FGFR kinase inhibitor; Pan-FGFR inhibitor; Selective FGFR inhibitor; FGFR pathway; FGFR signaling; Fibroblast growth factor; FGFR1; FGFR2; FGFR3; FGFR4; FGF; FGF19; FGF21; FGF23; FGFR mutation; FGFR gene fusion; FGFR gene translocation; FGFR genetic aberration; FGFR2 fusion; FGFR2 translocation; Phase 1 Clinical Trial; Phase I Clinical Trial; Clinical oncology; Tumor; Tumour; derazantinib; MK-2921
MeSH Terms: conditions — Liver Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma; Neoplasms | interventions — derazantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Low Dose Group (Experimental): Patients who received derazantinib orally at dose levels from 25 mg every other day (QOD) - 200 mg daily (QD) on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
  Interventions: Drug: Derazantinib low dose range
- Middle Dose Group (Experimental): Patients who received derazantinib orally at dose levels from 250 mg QD - 325 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
  Interventions: Drug: Derazantinib middle dose range
- High Dose Group (Experimental): Patients who received derazantinib orally at dose levels from 400 mg QD - 425 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
  Interventions: Drug: Derazantinib high dose range
- Expanded Cohort Group (Experimental): Patients who received derazantinib orally at the recommended phase 2 dose of 300 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
  Interventions: Drug: Derazantinib at recommended phase 2 dose (RP2D)

INTERVENTIONS:
Drug: Derazantinib low dose range — Derazantinib was administered orally at dose levels from 25 mg QOD - 200 mg QD on a 28-day schedule.
  Arms: Low Dose Group
Drug: Derazantinib middle dose range — Derazantinib was administered orally at dose levels from 250 mg QD - 325 mg QD on a 28-day schedule.
  Arms: Middle Dose Group
Drug: Derazantinib high dose range — Derazantinib was administered orally at dose levels from 400 mg QD - 425 mg QD on a 28-day schedule.
  Arms: High Dose Group
Drug: Derazantinib at recommended phase 2 dose (RP2D) — Derazantinib was administered orally at the recommended phase 2 dose of 300 mg QD on a 28-day schedule.
  Arms: Expanded Cohort Group

SUMMARY:
This was an open-label, Phase 1/2, dose escalation and signal finding study of derazantinib administered to patients with advanced solid tumors (Part 1; Dose Escalation/Food-effect Cohorts) or with advanced solid tumors with FGFR genetic aberrations, including iCCA with FGFR2 gene fusion (Part 2; Expanded Cohort, signal finding).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent granted
2. Men or women ≥18 years of age
3. Histologically or cytologically confirmed, locally advanced, inoperable, or metastatic solid tumors. Patients eligible for enrollment in the Expanded Cohort must have documented and/or confirmed FGFR genetic aberrations, including iCCA with FGFR2 gene fusion.
4. Failure to respond to standard therapy, or for whom standard therapy does not exist.
5. Evaluable or measurable disease
6. Archival and/or fresh biopsy tissue samples must be available prior to the first dose of the study drug
7. Life expectancy ≥ 12 weeks
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
9. Hemoglobin (Hgb) ≥ 9.0 g/dL
10. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
11. Platelet count ≥ 100 x 10^9/L
12. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (≤ 2 x ULN for patients with cholangiocarcinoma)
13. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 × ULN (≤ 5 x ULN for patients with liver metastases)
14. Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
15. Albumin ≥ 2.8 g/dL
16. INR 0.8 to ULN or ≤ 3 for patients receiving anticoagulant therapy
17. Men or women of child-producing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoid intercourse during the study and for 90 days after the last dose of study drug
18. Women of childbearing potential must have a negative serum pregnancy test during Screening Period and within 48 hours of the first dose of derazantinib.

Exclusion Criteria:

1. Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal, targeted therapy, or investigational agents within four weeks or five times of the drug half life, whichever is longer, of the first dose of derazantinib
2. Major surgery or radiation therapy within four weeks of the first dose of derazantinib
3. Previous treatment with FGFR inhibitors
4. History of allergic reactions attributed to compounds of similar chemical or biological composition as derazantinib
5. Unable or unwilling to swallow the complete daily dose of derazantinib
6. Clinically unstable central nervous system (CNS) metastasis
7. History of myocardial infarction (MI) or congestive heart failure defined as Class II to IV per the New York Heart Association classification within 6 months of the first dose of derazantinib (MI occurring >6 months of the first dose of derazantinib will be permitted)
8. Significant GI disorder(s) that could interfere with the absorption, metabolism, or excretion of derazantinib (e.g. Crohn's disease, ulcerative colitis, extensive gastric resection)
9. History and/or current evidence of clinically relevant ectopic mineralization/calcification
10. Previous malignancy within 2 years prior to the first dose of derazantinib, except curatively treated non-melanoma skin cancer, carcinoma in-situ of the breast or cervix, or superficial bladder tumors
11. Known human immunodeficiency virus (HIV) infection
12. Concurrent uncontrolled illness not related to cancer, including but not limited to:

    * Psychiatric illness/substance abuse/social situation that would limit compliance with study requirements.
    * Uncontrolled diabetes mellitus
13. Blood transfusion within 5 days of the blood draw being used to confirm eligibility
14. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica
Locations (12):
- United States (8):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - University of Washington, Seattle, Washington
- Italy (4):
  - Istituto Clinico Humanitas, Milan
  - Istituto Nazionale Tumori (National Cancer Institute), Milan
  - Instituto Oncologico Veneto, IRCCS, Padua
  - Azienda Ospedaliero-Universitaria Pisana - U.O. Oncologia Medica 2 Univ., Pisa

REFERENCES:
- [Result] Papadopoulos KP, El-Rayes BF, Tolcher AW, Patnaik A, Rasco DW, Harvey RD, LoRusso PM, Sachdev JC, Abbadessa G, Savage RE, Hall T, Schwartz B, Wang Y, Kazakin J, Shaib WL. A Phase 1 study of ARQ 087, an oral pan-FGFR inhibitor in patients with advanced solid tumours. Br J Cancer. 2017 Nov 21;117(11):1592-1599. doi: 10.1038/bjc.2017.330. Epub 2017 Oct 3. PMID 28972963
- [Result] Mazzaferro V, El-Rayes BF, Droz Dit Busset M, Cotsoglou C, Harris WP, Damjanov N, Masi G, Rimassa L, Personeni N, Braiteh F, Zagonel V, Papadopoulos KP, Hall T, Wang Y, Schwartz B, Kazakin J, Bhoori S, de Braud F, Shaib WL. Derazantinib (ARQ 087) in advanced or inoperable FGFR2 gene fusion-positive intrahepatic cholangiocarcinoma. Br J Cancer. 2019 Jan;120(2):165-171. doi: 10.1038/s41416-018-0334-0. Epub 2018 Nov 13. PMID 30420614
- [Derived] Hall TG, Yu Y, Eathiraj S, Wang Y, Savage RE, Lapierre JM, Schwartz B, Abbadessa G. Preclinical Activity of ARQ 087, a Novel Inhibitor Targeting FGFR Dysregulation. PLoS One. 2016 Sep 14;11(9):e0162594. doi: 10.1371/journal.pone.0162594. eCollection 2016. PMID 27627808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 12 study centers, 8 in the US and 4 in Italy. 119 subjects were recruited between December 2012 and January 2017.
Pre-assignment Details: A fresh core needle biopsy or fine needle aspiration could be collected during the screening period if archival tumor tissue biopsy samples were not available.
Groups:
- Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group: Subjects who received derazantinib orally at dose levels from 25 mg QOD - 200 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group: Subjects who received derazantinib orally at dose levels from 250 mg QD - 325 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 400 mg QOD - 425 mg QD - High Dose Group: Subjects who received derazantinib orally at dose levels from 400 mg QD - 425 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 300 mg QD - Expanded Cohort Group: Subjects who received derazantinib orally at the recommended phase 2 dose of 300 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
Period: Overall Study
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
Started | 29 | 13 | 19 | 58
Completed | 0 | 0 | 0 | 0
Not Completed | 29 | 13 | 19 | 58
Not completed — Adverse Event | 1 | 0 | 5 | 10
Not completed — Clinical Disease Progression | 6 | 4 | 1 | 13
Not completed — Physician Decision | 1 | 0 | 0 | 3
Not completed — Radiographic Disease Progression | 20 | 7 | 12 | 29
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Lack of clinical benefit | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population (patients who received any amount of derazantinib)
Groups:
- Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group: Patients who received derazantinib orally at dose levels from 25 mg QOD - 200 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 250 mg QOD - 325 mg QD - Middle Dose Group: Patients who received derazantinib orally at dose levels from 250 mg QD - 325 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 400 mg QOD - 425 mg QD - High Dose Group: Patients who received derazantinib orally at dose levels from 400 mg QD - 425 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Derazantinib 300 mg QD - Expanded Cohort Group: Patients who received derazantinib orally at the recommended phase 2 dose of 300 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
- Total: Total of all reporting groups
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD - Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group | Total
Number analyzed (Participants) | 29 | 13 | 19 | 58 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 4 | 8 | 35 | 66
  >=65 years | 10 | 9 | 11 | 23 | 53
Age, Continuous [Median (Full Range); unit: years] | 60 [34 to 72] | 67 [47 to 77] | 66 [41 to 78] | 60.5 [19 to 81] | 63 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 11 | 32 | 69
  Male | 12 | 4 | 8 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 2 | 9
  Not Hispanic or Latino | 26 | 12 | 16 | 56 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 3 | 9
  White | 24 | 11 | 16 | 54 | 105
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Drug-related Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events were graded for severity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. CTCAE is classifying AEs and their associated severity from Grade 1 (Mild AE), Grade 2 (Moderate AE), Grade 3 (Severe or medically significant but not immediately life-threatening), Grade 4 (Life-threatening consequences) to Grade 5 (Death related to AE)
Time Frame: Adverse events were collected and reported from the time of receiving first dose of derazantinib to the end of study assessment and follow-up period (30-day post-treatment)
Population: The safety population included all subjects who received at least one dose of derazantinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD - Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
Number analyzed (Participants) | 29 | 13 | 19 | 58
Participants
  TEAE Grade 1 | 3 | 1 | 1 | 11
  TEAE Grade 2 | 14 | 5 | 3 | 14
  TEAE Grade 3 | 9 | 6 | 13 | 24
  TEAE Grade 4 | 0 | 1 | 0 | 4
  TEAE Grade 5 | 2 | 0 | 2 | 5
  no TEAE | 1 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Patients With an Objective Tumor Response Per RECIST 1.1
Description: The number of patients with an objective tumor response, which included those with either a complete response (CR) or a partial response (PR) based on RECIST v1.1 guidelines which defines criteria for the radiological assessment in tumor response.
  The objective response rate (ORR) was defined as the proportion of patients with a CR or PR.
Time Frame: Assessments were performed at Baseline, and every 8 weeks during continuous drug administration until the End of Treatment visit (7 [+3] days after the last dose of derazantinib) or as otherwise clinically indicated.
Population: Evaluable Population: patients who received at least one cycle of study treatment and had at least one postbaseline tumor evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group: Patients who received derazantinib orally at dose levels from 250 mg QD - 325 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria.
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
Number analyzed (Participants) | 29 | 13 | 19 | 58
Participants | 0 | 0 | 1 | 5

3. Secondary Outcome: Proportion of Patients With Disease Control Per RECIST 1.1
Description: The number of patients with tumor disease control, which included those with either a complete or partial tumor response, or a stable disease (SD) based on RECIST v1.1 guidelines which defines criteria for the radiological assessment in tumor response. The disease control rate (DCR) was defined as the proportion of patients with CR, PR or SD.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Derazantinib 300 mg QD - Expanded Cohort Group: Patients who received derazantinib orally at the recommended phase 2 dose of 300 mg QD on a 28-day schedule until documented progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria .
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD - Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
Number analyzed (Participants) | 29 | 13 | 19 | 58
Participants | 8 | 4 | 7 | 32

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was calculated as the time from the date of first dose until documented radiographic disease progression or death from any cause, whichever occurred first. Disease progression is measured according to a specified radiologic increase in tumor size.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
Number analyzed (Participants) | 29 | 13 | 19 | 58
weeks | 8.3 [6.3 to 9.3] | 15.3 [6.7 to 22.1] | 8.1 [6.7 to 23.9] | 17.4 [7.9 to 24.9]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the first administration of study drug up to 30 days after the last study drug administration. The average period of time for AE data collection was 28 weeks.
Description: Adverse events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group | Derazantinib 300 mg QD - Expanded Cohort Group
All-Cause Mortality (participants affected / at risk) | 2/29 | 0/13 | 2/19 | 5/58
Serious Adverse Events (participants affected / at risk) | 9/29 | 2/13 | 6/19 | 16/58
Other Adverse Events (participants affected / at risk) | 28/29 | 13/13 | 19/19 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group (N=29) | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group (N=13) | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group (N=19) | Derazantinib 300 mg QD - Expanded Cohort Group (N=58)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord injury cervical (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Derazantinib 25 mg QOD - 200 mg QD - Low Dose Group (N=29) | Derazantinib 250 mg QOD - 325 mg QD -Middle Dose Group (N=13) | Derazantinib 400 mg QOD - 425 mg QD - High Dose Group (N=19) | Derazantinib 300 mg QD - Expanded Cohort Group (N=58)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 4 (6) | 17 (31)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 7 (10) | 10 (14) | 17 (30)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 2 (2) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 1 (1) | 4 (4) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 5 (6) | 2 (2) | 3 (3) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram QT interval abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity tests abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ichthyosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (12) | 3 (4) | 0 (0) | 10 (18)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Clumsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 5 (11) | 9 (15)
Dizziness postural (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 11 (14)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (5) | 12 (14)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (9)
Dry eye (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 7 (8)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (14)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (2) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 1 (1) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 8 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (5) | 7 (9) | 16 (20)
Diarrhoea (Gastrointestinal disorders) | 6 (11) | 5 (5) | 9 (10) | 17 (37)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (8) | 19 (23)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 6 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (18) | 8 (14) | 13 (15) | 27 (46)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (11) | 2 (5) | 7 (7) | 23 (48)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Micturition frequency decreased (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 11 (11)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (6) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 4 (4)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 3 (6) | 6 (8) | 13 (15)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (10) | 3 (4) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 2 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (4) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (26)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 18 (24) | 8 (14) | 11 (18) | 26 (40)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Performance status decreased (General disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 0 (0) | 1 (1) | 6 (9)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (5) | 3 (3) | 2 (3) | 2 (2)
Depression (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1) | 3 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT01752920/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT01752920/SAP_001.pdf